CLINICAL TRIAL: NCT05350332
Title: Characterizing the Effects of Lung Volume on Upper Airway Patency During Drug Induced Sleep Endoscopy in Patients With Obstructive Sleep Apnea
Brief Title: Effects of Lung Volume on Upper Airway Patency During Drug Induced Sleep Endoscopy
Acronym: DISE-Pulm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Lunair Medical (Industry)
Responsible Party: Principal Investigator, Jason Yu, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00003579
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Ventilators, Negative-Pressure; Respiratory Function Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Negative Pressure Ventilator (Experimental): Participants with obstructive sleep apnea (OSA) who are being evaluated for surgical treatment of their OSA and having a routine clinical DISE will have their lung volume increased with a non-invasive negative pressure ventilator. Participants will also have a pulmonary function test performed per routine clinical protocol, but for research purposes only (i.e., not part of usual care).
  Interventions: Device: Negative Pressure Ventilator; Device: Pulmonary Function Testing (PFT)
- Transcutaneous Phrenic Nerve Stimulation (Experimental): Participants with obstructive sleep apnea (OSA) who are being evaluated for surgical treatment of their OSA and having a routine clinical DISE will have their lung volume increased with transcutaneous phrenic nerve stimulation. Participants will also have a pulmonary function test performed per routine clinical protocol, but for research purposes only (i.e., not part of usual care).
  Interventions: Device: Pulmonary Function Testing (PFT); Device: Transcutaneous Phrenic Nerve Stimulation

INTERVENTIONS:
Device: Negative Pressure Ventilator — The negative pressure ventilator is an off-the-shelf FDA-approved device designed to treat respiratory patients with hypoventilation syndromes. This ventilator places the torso within a fixed container that is connected to a vacuum source, which inflates the lungs by pulling a negative pressure around the chest and abdomen. After the clinically routine DISE, a negative pressure ventilator will be placed on the participant's chest to increase lung volumes and the DISE evaluation will be repeated to observe changes.
  Other Names: cuirass ventilator; Hayek turtle shell; iron lung
  Arms: Negative Pressure Ventilator
Device: Pulmonary Function Testing (PFT) — PFT is a routine standardized clinical test evaluating lung function, consisting of two parts: spirometry and body plethysmography. In spirometry, participants breathe through a mouthpiece that measures airflow and volume to determine normal and maximal volume of inspiration/expiration. Body plethysmography is performed to calculate residual lung volumes. Participants enter in an enclosed chamber where they breathe through a mouthpiece. Changes in pressure in the sealed chamber during breathing are used to calculate the volume of air that remains in the lung after expiration. A MiniBox+ device may be used. The MiniBox+ device derives total lung capacity (TLC) during tidal breathing by the analysis of gas pressures and airflows immediately preceding and immediately following airway occlusions to calculate the same measures as conventional PFT analysis.
  Other Names: MiniBox+
Device: Transcutaneous Phrenic Nerve Stimulation — Phrenic nerve stimulation (PNS) will be performed transcutaneously using a commercially available and FDA approved peripheral neurostimulator. (Digitimer DS8R Bipolar Constant Current Stimulator). The neurostimulator consists of a stimulation generating box connected to electrodes that will be placed over the skin of the neck bilaterally over both phrenic nerves where an bipolar electric current will be used to stimulate the phrenic nerve leading to diaphragm contraction.
  Arms: Transcutaneous Phrenic Nerve Stimulation

SUMMARY:
Obstructive sleep apnea (OSA) is a disorder where a person has recurrent choking episodes during sleep. Surgery can treat OSA and drug induced sleep endoscopy (DISE) is a procedure that surgeons use to evaluate the throat while a person is sedated, mimicking sleep, to help determine if surgery might be effective. Lung volume can influence OSA severity but the relationship between lung function and throat collapse seen on DISE has not been well studied. This study aims to see if lung volume influences what is happening in the throat during DISE. Participants will be recruited from the sleep surgery clinic where they are being evaluated for surgery to treat their OSA. Participants will have a DISE that is performed as part of their routine surgical workup for treatment of OSA. Additionally, during the DISE, they will participate in one of two study groups. One group will have a negative pressure "turtle shell" ventilator placed over the participants chest during DISE to manipulate lung volumes to see if it can improve throat collapse. A second group will have electrodes placed over the neck to stimulate the phrenic nerve to contract the diaphragm to improve lung volumes to see if it can improve throat collapse. Both groups will also have a lung function test performed.The findings of this study will be important in improving pre-surgical evaluation of patients to better predict if surgery can help as well as potentially develop new surgical therapies for the treatment of OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disorder characterized by recurrent choking episodes during sleep. OSA affects over 25 million Americans and is associated with increased risks of hypertension, diabetes, cardiovascular disease, and stroke. The severity of OSA is measured by the number of complete or partial obstructive events per hour of sleep, and quantified for diagnostic and research purposes as the apnea-hypopnea index (AHI). Continuous positive airway pressure (CPAP) is the first line therapy for treating OSA, however, 20-40% of patients do not tolerate wearing a pressurized mask during sleep. Several surgeries can treat OSA, including pharyngeal soft tissue surgery, skeletal advancement surgery, and hypoglossal nerve stimulation which are deemed successful when surgery reduces the AHI to below 5 events per hour. Successful surgical treatment of OSA is highly variable with rates of success as low as 40% in early studies that looked at pharyngeal soft tissue surgery. Selecting OSA patients for surgery based on certain pathophysiologic characteristics has vastly improved surgical success rates, up to 60-80% depending on the surgery. However, the application of OSA pathophysiological assessment for surgical selection remains incomplete. This study will explore a wider range of pathophysiological factors to improve surgical outcomes and anticipate that further understanding of these relationships will support development of new surgical and non-surgical treatments for those who may not benefit from current treatment options.

Drug induced sleep endoscopy (DISE) is currently used to help determine appropriate patients for OSA surgery. During DISE, a fiber optic camera is placed through the nose into the throat to visualize airway collapse patterns during sedation mimicking natural sleep. The standardized method of describing airway collapse is known as the Velum, Oropharynx, Tongue Base, Epiglottis (VOTE) score which assesses the severity and pattern of collapse at four different anatomic sites of the upper airway. Previous studies have shown that airway collapse patterns visualized on DISE affect surgical outcomes.

Prior studies indicate that the phrenic nerve can be stimulated non-invasively to examine effects of diaphragmatic contraction on upper airway patency. Initial studies demonstrated that surface electrodes overlying the phrenic nerves in the lateral neck can be used to recruit the diaphragm and generate tidal breaths. Later studies demonstrated similar effects of transcutaneous stimulation with inductance coils on tidal airflow while modeling the effects of vigorous diaphragmatic contraction on pharyngeal patency. Finally, transcutaneous phrenic nerve stimulation has been applied during drug-induced sleep studies in patients to elucidate effects of lung volume on pharyngeal patency. This study demonstrated substantial reductions in upper airway obstruction in a dose-dependent fashion when phrenic nerve stimulation increased lung volume to varying levels. Of note, no untoward adverse events were noted in any of these prior studies. Taken together, these studies demonstrate that external transcutaneous stimulation is safe, can generate transient and sustained elevations in lung volume, and relieve upper airway obstruction in sedated individuals.

One overlooked pathophysiologic factor in the evaluation for OSA surgery is lung volume. Studies of lung physiology in OSA patients have found that lower functional residual capacity (FRC) and expiratory reserve volume (ERV) on pulmonary function testing, a commonly used procedure in pulmonary medicine, is associated with increased OSA severity. Experimental studies in OSA patients have shown that when negative pressure was used to expand the chest (e.g., iron lung) during sleep, the subsequent increased lung volume resulted in decreased upper airway collapsibility and reduced OSA severity. Transcutaneous phrenic nerve stimulation has also been applied during sedation studies in patients to elucidate effects of lung volume on pharyngeal patency demonstrating substantial reductions in upper airway obstruction in a dose-dependent fashion when phrenic nerve stimulation increased lung volume to varying levels. Despite this evidence, lung volume is not utilized as part of the evaluation for OSA surgery. The goal of this study is to determine if lung volume is useful in predicting surgical success and whether improving lung volumes via negative pressure ventilator or phrenic nerve stimulation can be used as an adjunctive therapy with surgery to treat OSA.

Patients will participate in DISE and be assigned either into a negative pressure ventilator or phrenic nerve stimulation cohort to evaluate each modality's effect on improving lung volume and altering upper airway collapsibility in DISE. Participants will also have a pulmonary function test to determine baseline lung volume measures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 yrs) willing and capable of providing informed consent
* Obstructive sleep apnea (AHI ≥ 5 events/hour)
* Must be willing and able to provide informed consent to participate in the study.
* Interested in surgical treatments of OSA and have consented for a DISE procedure as part of their routine clinical evaluation.

  * Patients are evaluated and cleared by anesthesia prior to the procedure.

Exclusion Criteria:

* No significant uncontrolled medical co-morbidities (e.g., uncontrolled hypertension, unstable angina, uncompensated heart failure or COPD).
* Any medical comorbidity that would prevent the patient from receiving anesthesia or having surgery
* Inability to tolerate negative pressure ventilator or perform PFT (i.e. claustrophobia)
* No incapacitating disability that interferes with execution of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Expiratory Reserve Volume (ERV) | During PFT
  ERV is the volume of extra air that can be forcefully breathed out after exhaling normally. ERV is impacted by body size and altitude and the normal range for adults is about 0.7 to 1.1 liters (L). ERV is obtained as part of the pulmonary function test.
Functional Residual Capacity (FRC) | During PFT
  FRC is the amount of air remaining in the lungs after a normal exhalation. FRC is impacted by body size and altitude and the normal volume for adults is about 1.8 to 2.4 L. FRC is obtained during the pulmonary function test and is the sum of residual volume (RV; the volume of air remaining after maximum exhalation) and ERV.
Change in VOTE Collapse Patterns - Degree of Obstruction | During clinical DISE and intervention DISE
  VOTE collapse patterns are obtained during the routine clinical DISE evaluation and during DISE with negative pressure ventilation. The VOTE classification codes degree of obstruction as 0 = no obstruction (no vibration), 1 = partial obstruction (vibration), and 2 = complete obstruction (collapse). Degree of obstruction is determined the velum, oropharynx lateral walls, tongue base, and epiglottis. The measurements obtained without and with negative pressure ventilation will be compared.
Change in VOTE Collapse Patterns - Configuration of Obstruction | During clinical DISE and intervention DISE
  VOTE collapse patterns are obtained during the routine clinical DISE evaluation and during DISE with negative pressure ventilation. The VOTE classification codes configuration of obstruction for structures with a degree of obstruction greater than 0. The configuration of obstruction is categorized as anteroposterior (anterior structures moving posteriorly against pharyngeal wall), lateral (lateral structures moving towards airway center), or concentric (both anteroposterior and lateral movements). The measurements obtained without and with negative pressure ventilation will be compared.
Change in Critical Closing Pressure (Pcrit) | During clinical DISE and intervention DISE
  Critical closing pressures are obtained during the routine clinical DISE evaluation and during DISE with negative pressure ventilation. Pcrit assessed pharyngeal collapsibility and is measured as centimeters of water (cm H2O). A Pcrit of less than -10 cm H2O indicates normal breathing. Patients with a Pcrit around -6cm H2O tend to snore but not have OSA. A Pcrit around or greater than 0 cm H2O is seen with obstructive sleep apnea.The measurements obtained without and with negative pressure ventilation will be compared.
Change in Pharyngeal Opening Pressures | During clinical DISE and intervention DISE
  Pharyngeal opening pressures are obtained during the routine clinical DISE evaluation and during DISE with negative pressure ventilation. Opening pressures are obtained using a positive airway pressure (PAP) titration device. Pharyngeal opening pressures are defined as the minimally effective positive airway pressure that results in non-flow limited breathing. This is measured in cm H2O and ranges from 0 to 25 cm H2O, with 25 cm H2O being the maximum pressure the PAP machine is capable of generating. The measurements obtained without and with negative pressure ventilation will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Yu, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial after deidentification will be available to share to researchers who provide a methodologically sound proposal. Sharing will be available immediately following publication with no end date.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposal should be directed to jason.lee.yu@emory.edu.

REFERENCES:
- [Background] Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000 May 11;342(19):1378-84. doi: 10.1056/NEJM200005113421901. PMID 10805822
- [Background] Punjabi NM, Shahar E, Redline S, Gottlieb DJ, Givelber R, Resnick HE; Sleep Heart Health Study Investigators. Sleep-disordered breathing, glucose intolerance, and insulin resistance: the Sleep Heart Health Study. Am J Epidemiol. 2004 Sep 15;160(6):521-30. doi: 10.1093/aje/kwh261. PMID 15353412
- [Background] Drager LF, Bortolotto LA, Lorenzi MC, Figueiredo AC, Krieger EM, Lorenzi-Filho G. Early signs of atherosclerosis in obstructive sleep apnea. Am J Respir Crit Care Med. 2005 Sep 1;172(5):613-8. doi: 10.1164/rccm.200503-340OC. Epub 2005 May 18. PMID 15901608
- [Background] Yaggi HK, Concato J, Kernan WN, Lichtman JH, Brass LM, Mohsenin V. Obstructive sleep apnea as a risk factor for stroke and death. N Engl J Med. 2005 Nov 10;353(19):2034-41. doi: 10.1056/NEJMoa043104. PMID 16282178
- [Background] Punjabi NM. The epidemiology of adult obstructive sleep apnea. Proc Am Thorac Soc. 2008 Feb 15;5(2):136-43. doi: 10.1513/pats.200709-155MG. PMID 18250205
- [Background] Iber, Conrad, Ancoli-Israel, Sonia, Chesson, Andrew L, Quan, Stuart F. The AASM manual for the scoring of sleep and associated events: rules, terminology and technical specifications. Am Acad Sleep Med Westchest IL. 2007;1.
- [Background] Richards D, Bartlett DJ, Wong K, Malouff J, Grunstein RR. Increased adherence to CPAP with a group cognitive behavioral treatment intervention: a randomized trial. Sleep. 2007 May;30(5):635-40. doi: 10.1093/sleep/30.5.635. PMID 17552379
- [Background] Weaver TE, Grunstein RR. Adherence to continuous positive airway pressure therapy: the challenge to effective treatment. Proc Am Thorac Soc. 2008 Feb 15;5(2):173-8. doi: 10.1513/pats.200708-119MG. PMID 18250209
- [Background] Veasey SC, Rosen IM. Obstructive Sleep Apnea in Adults. N Engl J Med. 2019 Apr 11;380(15):1442-1449. doi: 10.1056/NEJMcp1816152. No abstract available. PMID 30970189
- [Background] Pepin JL, Woehrle H, Liu D, Shao S, Armitstead JP, Cistulli PA, Benjafield AV, Malhotra A. Adherence to Positive Airway Therapy After Switching From CPAP to ASV: A Big Data Analysis. J Clin Sleep Med. 2018 Jan 15;14(1):57-63. doi: 10.5664/jcsm.6880. PMID 29198291
- [Background] Bakker JP, Weaver TE, Parthasarathy S, Aloia MS. Adherence to CPAP: What Should We Be Aiming For, and How Can We Get There? Chest. 2019 Jun;155(6):1272-1287. doi: 10.1016/j.chest.2019.01.012. Epub 2019 Jan 23. PMID 30684472
- [Background] Verse T, Kroker BA, Pirsig W, Brosch S. Tonsillectomy as a treatment of obstructive sleep apnea in adults with tonsillar hypertrophy. Laryngoscope. 2000 Sep;110(9):1556-9. doi: 10.1097/00005537-200009000-00029. PMID 10983961
- [Background] Series F, Cormier Y, Lampron N, La Forge J. Increasing the functional residual capacity may reverse obstructive sleep apnea. Sleep. 1988 Aug;11(4):349-53. PMID 2974620
- [Background] Heinzer RC, Stanchina ML, Malhotra A, Jordan AS, Patel SR, Lo YL, Wellman A, Schory K, Dover L, White DP. Effect of increased lung volume on sleep disordered breathing in patients with sleep apnoea. Thorax. 2006 May;61(5):435-9. doi: 10.1136/thx.2005.052084. Epub 2006 Feb 20. PMID 16490766
- [Background] Owens RL, Malhotra A, Eckert DJ, White DP, Jordan AS. The influence of end-expiratory lung volume on measurements of pharyngeal collapsibility. J Appl Physiol (1985). 2010 Feb;108(2):445-51. doi: 10.1152/japplphysiol.00755.2009. Epub 2009 Nov 25. PMID 19940097
- [Derived] Chan TG, Plageman J, Yu JL. The Repeatability of Pharyngeal Opening Pressure Under Drug-Induced Sleep Endoscopy. Otolaryngol Head Neck Surg. 2024 Jul;171(1):295-302. doi: 10.1002/ohn.730. Epub 2024 Apr 12. PMID 38606621